CLINICAL TRIAL: NCT06789939
Title: Impact of Interprofessional Education in Multidisciplinary Primary Care Centres on Collaborative Competency of Healthcare Students - Quasi-experimental Study
Brief Title: Impact of IPE in Multidisciplinary Primary Care Centres on Collaborative Competency of Healthcare Students (FLIRT-MSP)
Acronym: FLIRT-MSP
Status: Not yet recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC22_8980_FLIRT-MSP
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Interprofessional Education
Keywords: Primary Health Care; Interprofessional collaboration; Self evaluation program; Students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MPCC participating in intervention group: * MPCC signatories to the interprofessional conventional agreement with the French national health insurance system
  * volunteer to take part in the FLIRT MSP Study
  * volunteer to form an interprofessional training team
  * MPCC with GPs who are habilitated to supervise internship family medicine students
  * MPCC volunteer to receive healthcare students from different professions including at least one GP intern.
  Interventions: Other: Train the trainer program for MPCC professionals
- MPCC participating in control group: * MPCC signatories to the interprofessional conventional agreement with the French national health insurance system
  * volunteer to take part in the FLIRT MSP Study
  * MPCC with GPs who receive internship family medicine students
  * MPCC volunteer to receive healthcare students from different professions including at least one GP intern.

INTERVENTIONS:
Other: Train the trainer program for MPCC professionals — The intervention will consist on a train the trainer program. 3 professionals from each MPCC will be trained by an educational team. They will then have to implement an IPEP (knowledge of the MPCC, participation in interprofessional MPCC activities, etc.) for students on placement in their MPCC.
  Groups: MPCC participating in intervention group

SUMMARY:
The aim of our study is to evaluate the impact of interprofessional education program (IPEP) for healthcare students in clinical placement in MPCC on interprofessional collaboration (IPC), comparing the acquisition of interprofessional collaboration skills in students receiving IPEP during their MPCC placement with those in their MPCC placements without this IPEP.

The IPEP will be delivered by trainers (health professionnals from the MPCC) who receive a train the trainer program.

DETAILED DESCRIPTION:
For the intervention group, 12 MPCC will be recruited. 3 professionals from each MPCC will be trained and will be responsible for implementing the IPEP for their students.

For the control group, 12 MPCC will be recruited. Students will carry out their clinical placement as usual.

Study method : A multimodal study with a quasi experimental multisite study before and after the IPEP and a qualitative study to explore students' perceptions of the IPC will be conducted.

ELIGIBILITY:
Inclusion Criteria :

MPCC signatories to the interprofessional conventional agreement with the French national health insurance system.

Volunteer to take part in the FLIRT MSP Study. MPCC with GPs who are habilitated to supervise internship family medicine students.

MPCC volunteer to receive healthcare students from different professions including at least one GP intern.

Volunteer to form an interprofessional training team.

Exclusion Criteria:

MPCC who are unable to form an internship training team or to commit to IPE as stipulated in the protocol will not be included in the MSP intervention group.

For the qualitative study, students who do not volunteer or are unavailable for interview will not be included in the FLIRT qualitative component.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants in this study will be :
  * General medicine internship students in Level 1 (7th year) who complete 6-month internships with GPs.
  * Midwifery students doing internships with independent midwives.
  * Occupational therapy students who do internships with occupational therapists in private practice.
  * Pharmacy students (6th year), who complete 6-month internships in community pharmacies.
  * Other students doing clinical placements in MPCCs. A minimum of 48 students are expected to complete internships in MSPs as part of the intervention group.
  An equivalent number of at least 48 MSP students in the control group is planned.
  Students will be informed of the FLIRT study (intervention and control arms) when they receive the questionnaire, and will agree to take part.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of changes in student scores on the ICCAS (Interprofessional Collaborative Competency Attainment Survey) before and after the MPCC placement in the intervention and control groups. | 18 months

SECONDARY OUTCOMES:
Comparison of changes in student scores on the ICCAS for each of the 6 IPC dimensions in the intervention and control groups | 18 months
Comparison of changes in student scores on the ICCAS for each healthcare profession in the intervention and the control groups | 18 months
Analysis of the experience and feelings of students who have benefited from the IPEP on placement concerning their training and their vision of interprofessional collaboration (qualitative study). | 24 months
  The aim will be to understand how the placement changed their view of IPC, how they integrated into the MPCC, how they perceived interprofessional work and how they perceived their professional role within an MPCC.
Analysis of the feelings of students who did not benefit from IPEP on placement in relation to their education and their view of interprofessional collaboration (qualitative study). | 24 months
  The aim will be to understand how the placement changed their view of IPC, how they integrated into the MPCC, how they perceived interprofessional work and how they perceived their professional role within an MPCC.

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers

REFERENCES:
- [Background] Miselis HH, Zawacki S, White S, Yinusa-Nyahkoon L, Mostow C, Furlong J, Mott KK, Kumar A, Winter MR, Berklein F, Jack B. Interprofessional education in the clinical learning environment: a mixed-methods evaluation of a longitudinal experience in the primary care setting. J Interprof Care. 2022 Nov-Dec;36(6):845-855. doi: 10.1080/13561820.2022.2025768. Epub 2022 Feb 2. PMID 35109762
- [Background] Reeves S, Zwarenstein M, Goldman J, Barr H, Freeth D, Koppel I, Hammick M. The effectiveness of interprofessional education: key findings from a new systematic review. J Interprof Care. 2010 May;24(3):230-41. doi: 10.3109/13561820903163405. PMID 20178425
- [Background] Poitras ME, Couturier Y, Doucet E, T Vaillancourt V, Poirier MD, Gauthier G, Hudon C, Delli-Colli N, Gagnon D, Careau E, Duhoux A, Gaboury I, Charif AB, Ashcroft R, Lukewich J, Ramond-Roquin A, Masse S. Co-design, implementation, and evaluation of an expanded train-the-trainer strategy to support the sustainability of evidence-based practice guides for registered nurses and social workers in primary care clinics: a developmental evaluation protocol. BMC Prim Care. 2022 Apr 18;23(1):84. doi: 10.1186/s12875-022-01684-0. PMID 35436845